CLINICAL TRIAL: NCT01568879
Title: Evaluating the Effectiveness of a Chronic Disease Management Program for Gout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN-11RGold-02-H
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Recurrent or Tophaceous Gout
Keywords: Recurrent gout; Tophaceous gout; Gout flares; Arthritis; Joint Diseases; Rheumatic Diseases
MeSH Terms: conditions — Recurrence; Gout; Arthritis; Joint Diseases; Rheumatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gout Chronic Disease Management Program (Experimental)
  Interventions: Other: Gout Disease Management Program
- Usual Care (Active Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — The control group will receive care from their primary care physician that reflects the actual current care received by KPNC patients, but will not receive any treatment recommendations from the study protocol. The control subject will have regular monitoring of serum uric acid levels and will be provided with educational material and dietary counseling.
  Arms: Usual Care
Other: Gout Disease Management Program — The experimental group will utilize standard guidelines for the initiation of uric acid lowering treatments, and approved medications. The study protocol treatments include medication management, dietary guidelines, and basic educational materials on gout and its management. No non-formulary medications or devices will be used. The experimental procedure to be tested is the use of a structured protocol to manage and monitor standard treatments.
  Arms: Gout Chronic Disease Management Program

SUMMARY:
The aim of this study is to test the effectiveness of a pharmacist-staffed, protocol-based chronic disease management program compared to patients receiving usual care in achieving a target serum uric acid level in patients with recurrent gout.

DETAILED DESCRIPTION:
Gout is a chronic condition with intermittent symptoms and should be managed through an outcome-based disease management approach. Unlike other common chronic conditions, strategies for population management in gout patients have not been tested. The study will identify adult members of Kaiser Permanente (KP) Northern California with a diagnosis of gout and 3 or more outpatient or Emergency Department visits for gout over a 1-year period preceding study enrollment. These patients will be randomized to either an active management group, or to usual care. The participants will be enrolled and followed over a period of 26 weeks. The primary outcome to be measured will be the attainment and maintenance of a uric acid lowering regimen targeted to achieve serum uric acid level of 6.0 mg/dl or less. The treatment protocol will use standard treatment guidelines to lower and maintain uric acid levels to less than or equal to 6.0 mg/dl (or maximum doses of uric acid lowering medications) and provide patient education and dietary counseling. Monitoring and medication management will be carried out by a licensed clinical pharmacist under the supervision of an experienced rheumatologist. Control subjects will have regular monitoring of serum uric acid levels and will be provided with educational material and dietary counseling, but otherwise receive usual care. The demonstration that a chronic disease management approach to gout care can improve the health and reduce morbidity in patients with gout may illuminate a simple path towards improved quality of life and reduced morbidity in this growing population of patients.

ELIGIBILITY:
Inclusion Criteria:

Three or more outpatient/ED visits in a 24-month period prior to selection for study with one of these primary visit diagnoses:

* Gouty arthropathy
* Gout, unspecified
* Gout with other specified manifestations
* Tophaceous gout of ear (274.81) or other sites
* Gouty nephropathy

At least 2 years of continuous Kaiser Foundation Hospital Plan membership

Baseline uric acid level above 7.0mg/dl

Exclusion Criteria:

* Current cancer diagnosis with active treatment
* End stage renal disease
* Pregnant or lactating
* Patients with a diagnosis of dementia
* Terminally ill patients

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Serum Uric Acid Level | change from baseline at 6 months follow up
  attainment and maintenance of a serum uric acid level of 6.0 mg/dl or less. The outcome will be considered positive if that level is attained and the 6 month follow up value remains at the target level.

SECONDARY OUTCOMES:
Serum Creatinine | 0, 12, and 26 weeks
  Change in Serum Creatinine
Serum Alanine Aminotransferase (ALT) | 0, 12, and 26 weeks
  Change in serum ALT (a measure of potential toxicity)
Gout flares | 0, 12, and 26 weeks
  Number of gout flares

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldfien, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Northern California Medical Facilities, All KPNC Facilities, California, United States